CLINICAL TRIAL: NCT06267443
Title: Comparison of Two Different Techniques for Postoperative Analgesia in Cardiopulmonary Bypass Surgeries: Erector Spinae Plane Block or Parasternal Block Plus Chest Tube Wound Infiltration
Brief Title: Erector Spina Block or Parasternal Block Plus Chest Tube Wound Infiltration for Cardiac Surgeries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ayse Ulgey, PROFESSOR DR, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/337
Record Dates: First submitted 2023-12-25; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Postoperative Pain; Postoperative Atelectasis; Analgesia
Keywords: CPBGS; postop analgesia; ESPB; parasternal block; local anesthetic
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Active Comparator): in this group erector spina plane block will be performed before surgery for post operative analgesia
  Interventions: Procedure: Comparison of erector spina plane block, parasternal block plus local infiltration to the tube sides for postoperative analgesia
- Group 2 (Active Comparator): in this group after endotracheal intubation bilateral parasternal block will be performed and to the chest tube sides local anesthetic infiltration will be performed
  Interventions: Procedure: Comparison of erector spina plane block, parasternal block plus local infiltration to the tube sides for postoperative analgesia

INTERVENTIONS:
Procedure: Comparison of erector spina plane block, parasternal block plus local infiltration to the tube sides for postoperative analgesia — Group 1: erector spina plane block: With USG guidance at the thoracal level of 4-5, with 20ml 2.5% bupivacaine ESPB will be performed. after surgery in the ICU pain score and atelectasia will be evaluated.
  Group 2: With USG guidance parasternal block will be performed after intubation bilaterally with 10 ml 0.25% bupivacaine each side. at the end of the surgery infiltration of chest tube sides will be performed with 10 ml 2.5% bupivacain.

SUMMARY:
Pain management is important after coronary artery bypass graft (CABG) surgery. Intravenous morphine is the gold standard for pain relief, but its sedation, cough suppression and decreased bowel movements limit its use. Analgesia with regional methods after surgery provides effective analgesia by reducing morphine consumption. In this study we have planned to compare the erector spina plane block with parasternal block +local infiltration to chest tube areas.

DETAILED DESCRIPTION:
Patients who will undergo open heart surgery will be included in this study. Pain management is important after coronary artery bypass graft (CABG) surgery. Poorly controlled postoperative pain can trigger myocardial ischemia, increase catecholamine levels, result in increased complications such as stroke and bleeding, and increase the risk of pneumonia. Intravenous morphine is the gold standard for pain relief, but its sedation, cough suppression and decreased bowel movements limit its use. For this reason, regional methods are gaining importance in pain treatment. After cardiac surgery. Both sternotomy and bilateral chest tubes are the most painful interventions during cardiac surgeries. Parasternal block can be a good alternative in the treatment of pain in CABG surgeries. In parasternal application, the aim is to anesthetize the nerves innervating the sternum between the pectoral muscle and the intercostal muscle by holding the probe in the parasagittal plane on the lateral side of the sternum under USG guidance. Patients who will undergo open heart surgery will be included in this study. The patients will be divided into two groups, and in Group 1, before general anesthesia is given, bilateral ESPB will be performed at the 4-6th thoracic level in the prone position, and then routine general anesthesia will be performed (at this stage, the patients will be given sedation to prevent them from feeling pain). After endotracheal intubation, in Group 2, a parasternal block will be performed from the lateral sternum. At the end of the surgery, local anesthetic infiltration will be perform to the tube sites. General anesthesia and surgical procedures will be performed routinely in both groups. In the intensive care unit patients will be monitored for pain levels, intubation duration, whether there is atelectasis in the lungs, and the need for reintubation. Pain assessment will be evaluated with the behavioral pain score while the patients are intubated and with the visual pain scale after extubation. Whether atelectasis has developed will be evaluated with ultrasonography at the 12th and 24th hours postoperatively

ELIGIBILITY:
Inclusion Criteria:

1. Patients who will undergo open heart surgery
2. Patients who agreed to participate in the study-

Exclusion Criteria:

1. Patients who do not agree to participate in the study
2. Patients with chronic lung disease
3. Patients with D. Mellitus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
postoperative analgesia | 24 hours after after surgery
  postoperatively in the intensive care unit during mechanical ventilation behavioral pain, score, after extubation visüel analog scala will be used to measure postoperative pain of the patients. during mechanical ventilation every 2 hours after extübation 2., 4., 6., 8., 12., 24. hours
postoperative atelectasia | 24 hours after after surgery
  postoperatively at the 12. th and 24.th hours with ultrasonography the patients lungs will be sreened for atelectasis

SECONDARY OUTCOMES:
postoperative mechanical ventilation duration | 24 hours after after surgery
  in the intensive care unit time to endotracheal extubation will be recorded